CLINICAL TRIAL: NCT06800534
Title: Perineal and Abdominal Reconstruction: a Comparison of Reconstructive Methodologies
Acronym: PLAST-GEN-1
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PLAST-GEN-1
Record Dates: First submitted 2025-01-09; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The different reconstructive methods (V-Y flap, lotus flap, gracilis muscle flap, TRAM flap) will be compared with the complications that occurred following the surgery, so as to define which reconstructive methods have led to fewer complications and in which categories of patients.

DETAILED DESCRIPTION:
he study is of a non-interventional observational nature. It involves the collection of patient data in pseudonymous form from preoperative and postoperative assessments in accordance with daily clinical practice and normally performed for proper patient management.

The data recorded in the study are obtained from the medical records of patients who are normally accessed by the doctors of the operating unit during daily practice.

After having performed a meticulous collection of the basic data of the patients (gender, age, remote pathological history, recent pathological history, type of demolitive and reconstructive surgery performed), the different reconstructive methods (V-Y flap, lotus flap, gracilis muscle flap, TRAM flap) will be compared with the complications that occurred following the surgery, so as to define which reconstructive methods have led to fewer complications and in which categories of patients.

The complications are assessed through the retrospective analysis of the outpatient reports that are normally drawn up during the usual follow-up outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pelvic-perineal amputations for oncological disease or chronic inflammatory diseases whose surgical treatment required the collaboration of the plastic surgeon
* Patients with complications in the abdominal or pelvic-perineal region of surgical relevance and requiring reconstruction (enteric fistulas, abdominal wall defects)
* Age greater than or equal to 18 years
* Acquisition of written informed consent

Exclusion Criteria:

* Incomplete or missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population consists of subjects affected by rectal or vulvar neoplasia or chronic inflammatory bowel disease and subjected to demolition surgery at the General Surgery Unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna and related reconstruction (performed by the Plastic Surgery Unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna) in the period between 01/01/2011 and 31/12/2021.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success | From the first patient enrolled to the 50th patient, an average of 2 years
  Technical success is assessed by the number of reinterventions after 1 year from the treatment and the number of major complications.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pignatti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy